CLINICAL TRIAL: NCT01495273
Title: Adaptation of Nerve Stimulation Technology to Aid Transtracheal Needle Insertion and Injection
Brief Title: Electrically Guided Needle Insertion: Transtracheal Injection
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never started, no subjects enrolled
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00026789
Record Dates: First submitted 2011-11-17; First posted 2011-12-20 (Estimated); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Transtracheal Injection; Fibreoptic Intubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nerve stimulator (Experimental): Experimental group; will undergo transtracheal injection with needle connected to nerve stimulator.
  Interventions: Procedure: Transtracheal injection
- Standard needle/syringe (Active Comparator): Control group; will undergo transtracheal injection with standard needle/syringe assembly.
  Interventions: Procedure: Transtracheal injection

INTERVENTIONS:
Procedure: Transtracheal injection — Experimental group will undergo transtracheal injection using needle connected to a nerve stimulator device.
  Arms: Nerve stimulator
Procedure: Transtracheal injection — Control group will undergo transtracheal injection with a standard needle/syringe assembly.
  Arms: Standard needle/syringe

SUMMARY:
Various medical procedures require different objects to be inserted into the airway; for example, a bronchoscope - a fibreoptic camera device - can be guided down the windpipe to gain real-time images of the airway. Since inserting objects down the throat is uncomfortable for most patients, doctors have several options, one of which is putting the patient to sleep using general anesthetic before inserting something into the windpipe. This may not always be the best option, especially in cases where the patient needs to be awake during the procedure. In these cases, the doctor may 'freeze' the windpipe before inserting a scope or a tube into the airway. For this, the doctor inserts a needle through the front of the neck and injects local anesthetic. Inserting a needle into the windpipe comes with some risks to the patient, and the doctor wants to avoid puncturing nearby structures, such as arteries, veins, and the esophagus. The investigators have come up with a new method for accurately guiding a needle into the airway that will alert the user when they have successfully placed the needle tip in the windpipe. The investigators hypothesize that this new method will prove to be beneficial to clinicians and emergency medical personnel who need a fast, easy, and reliable way to insert a needle into the airway.

DETAILED DESCRIPTION:
Background and rationale

The trachea can be anesthetized by several different methods, one of which is transtracheal injection of a local anesthetic such as lidocaine. This technique is performed to prepare a patient for a variety of procedures, including awake fibreoptic intubation and cricothyroidotomy. Tracheal anesthesia is performed by first identifying the cricothyroid ligament; this structure is generally located by placing one finger on the thyroid cartilage and another on the cricoid cartilage. Approximately 4-6 mL of local anesthetic is delivered through a small needle or an intravenous catheter inserted in the neck midline. Anesthesia occurs quickly and permits the patient to be awake and aware during the procedures that follow.

Insertion of a needle into the trachea is not without risk to the patient. Several complicating factors affect the success rate of tracheal needle insertion, and in emergency situations where oxygen must be delivered through the insertion site, as in cricothyroidotomy, accurate needle insertion can mean the difference between life and death for the patient. One complicating factor in this procedure is that the thyroid cartilage and the cricoid cartilage can be difficult to identify, especially in obese people. Needle insertion is made more complicated due to the anatomy surrounding the cricothyroid membrane: the carotid artery and jugular vein lie laterally to the membrane, the cricothyroid artery is located superiorly and laterally, and the highly vascularized thyroid gland is located inferiorly. Intravascular injection of anesthetic can lead to a seizure, and inaccurate injection could lead to anesthesia of surrounding nerves. There is also a risk of puncturing through the posterior wall of the trachea, which may cause esophageal perforation.

Given these complications, a quick and easy method of ensuring accurate tracheal needle insertion, while avoiding damage to surrounding tissues, would greatly benefit clinicians and could potentially save lives in emergency situations. We wish to evaluate a simple technique to guide a needle tip into the trachea that mitigates the risks of conventional methods of needle insertion. We will use nerve stimulation equipment to aid in the guidance and placement of a needle tip into the tracheal lumen, which we predict will be faster and more accurate than current conventional methods. The nerve stimulation technology can alert the user to the exact moment the needle tip is suspended in the trachea and also alerts the user to when the needle tip is in contact with body tissue, avoiding accidental puncture of the lateral and posterior tracheal walls. We believe that this method of electrically-guided needle insertion will be a significant improvement over current methods of percutaneous needle insertion and transtracheal injection.

Study objective To assess the value of nerve stimulation equipment for guidance and placement of a needle-catheter assembly for transtracheal injection.

Hypothesis Nerve stimulation equipment will help the physician guide and insert the needle tip into the tracheal lumen with more accuracy than conventional techniques.

Study Design This is a prospective, descriptive, interventional study.

Study Procedures This study will involve recruiting consenting patients undergoing procedures that require awake fibreoptic intubation following transtracheal injection of local anesthetic. We intend to recruit 30 patients, who will be randomized into two groups, one (experimental) that will undergo transtracheal injection using a needle connected to a nerve stimulation device, and another (control) that will receive tracheal anesthetic using standard, conventional needle insertion and injection technique.

Patients will lay supine with the head and neck in a neutral position on one pillow. The physician will locate the cricothyroid ligament, through which the needle-catheter assembly will be inserted. In the experimental group, a 21G 64 mm insulated needle with an 18G catheter assembly (MultiSet, Pajunk, Germany) and a commonly used nerve stimulator (HNS 12, B.Braun, Germany) will be used to access the airway (this nerve stimulator device has been approved for use on live patients in Canada and is a common piece of equipment in operating rooms). The nerve stimulator will be connected to a current meter, and a ground electrode will be attached to the body. When the needle tip is in contact with body tissue (i.e., tracheal wall), the electrical circuit will be closed, producing a reading of 1.0 mA on the current reader. Suspension of the needle tip in the airway will interrupt the circuit, producing a reading of 0.0 mA. In addition, an audible signal built into the nerve stimulator will alert the user to a change in current, warning that the needle tip has advanced too far and is in contact with the posterior or lateral tracheal wall. Once the physician has successfully inserted the needle tip into the tracheal lumen, the needle will be withdrawn and 4-6 mL lidocaine (2-4%) will be delivered through the catheter, anesthetizing the airway. Once the airway is anesthetized, a bronchoscope can be guided down the trachea. The control group will undergo an identical procedure, except that no nerve stimulator will be connected to the needle.

For each patient, the physician performing the transtracheal injection will document their opinion of each needle insertion and injection, but no personal information about the patient will be recorded at this time. For both the experimental and control groups, study investigators will collect data documenting the time needed for each needle insertion and the success of each attempt. These data will be statistically analyzed to determine the value of the nerve stimulator-guided technique over the conventional technique.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years of age or older) patients who have provided informed consent.
* Require awake fibreoptic intubation.

Exclusion Criteria:

* Inability to consent due to language barrier or incapacity to consent.
* Known upper airway pathologies
* Known oro-pharyngeal or laryngeal disease, including any swelling, tumour, or infection.
* Previous radiotherapy or operations on the neck.
* Cervical spine fractures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-05 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Needle tip placement in tracheal lumen | From positioning of the patient to anesthesia of the trachea; approximately 10 minutes
  After injection of local anesthetic into the skin of the neck, a needle connected to a syringe containing 4-6 mL 2-4% lidocaine will be inserted through the cricothyroid membrane into the tracheal lumen. Success will be recorded as accurate puncture of the cricothyroid membrane and trachea and injection of lidocaine into the tracheal lumen.

CONTACTS AND LOCATIONS:
Overall Officials: Ban Tsui, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada